CLINICAL TRIAL: NCT03746444
Title: Comparison of Effects of Combined Spinoepidural and General Anesthesia Effects on Incidence of Postoperative Complications Following Total Knee Arthroplasty
Brief Title: Postoperative Complications Following Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Perihan Ekmekçi, Primary Investigator, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1001201311
Record Dates: First submitted 2018-10-15; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: total knee arthroplasty; general anesthesia; neuraxial anesthesia; complications
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General Anesthesia (Active Comparator): The patients in this group will undergo unilateral total knee arthroplasty under general anesthesia. Following vascular access and monitorization (non-invasive blood pressure, saturation, electrocardiography).
  Epidural chateterisation will be performed and test dose will be applied. Induction will be carried out using propofol (3mg/kg), fentanyl (1cmg/kg) and rocuronium (0.6 mg/kg). Maintenance will be carried out using sevoflurane (%2-3) and 50-50% mixture of nitrous oxide and oxygen. Epidural analgesia will be initiated after the end surgery.
  Interventions: Other: General Anesthesia
- Regional Anesthesia (Active Comparator): The patients in this group will undergo unilateral total knee arthroplasty under combined spinoedpidural anesthesia . Following vascular access and monitorization (noninvasive blood pressure, oxygen saturation and electrocardiography), spinal anesthesia will be performed using 12,5 mg marcaine given to the subarachnoid space and epidural analgesia will be initiated at the end of surgery following negative test dose. The patients will be given nasal oxygen supplementation.
  Interventions: Other: Regional Anesthesia

INTERVENTIONS:
Other: General Anesthesia — The patients in general anesthesia group will undergo general anesthesia
  Arms: General Anesthesia
Other: Regional Anesthesia — The patients in Group R will be given combined spinoepidural anesthesia
  Arms: Regional Anesthesia

SUMMARY:
The aim of this study is to investigate the effect of combined spinoepidural and general anesthesia on the incidence of postoperative complications following total knee arthroplasty

DETAILED DESCRIPTION:
Total knee arthroplasty is known to cause complications (pulmonary thromboembolism, acute kidney injury, arryhthmias and infection). The investigators aimed to study the effects of two different anesthesia techniques, i.e. combined spinoepidural anesthesia and general anesthesia on the incidence of postoperative complications such as arrhythmia, pulmonary thrombeoembolism, infection, acute kidney injury and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective unilateral total knee arthroplasty

Exclusion Criteria:

* Patient refusal
* Scheduled for bilateral or unilateral unicondylar knee arthroplasty
* Known history of allergy to drugs used in the study
* Severe systemic disease
* Morbid obesity (BMI>30)
* History of renal dysfunction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2018-12-20 (Estimated); Study Completion 2018-12-25 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | Postoperative first day
  Number of participants with new onset acute kidney injury
Acute Kidney Injury | Postoperative sixth week
  Number of participants with new onset acute kidney injury
Pulmonary Thromboembolism | Postoperative first day
  Number of participants with new onset pulmonary thromboembolism
Pulmonary Thromboembolism | Postoperative sixth week
  Number of participants with new onset pulmonary thromboembolism
Infection | Postoperative first day
  Number of participants with new onset infection
Infection | Postoperative sixth week
  Number of participants with new onset infection
Arryhthmia | Postoperative first day
  Number of participants with new onset arryhthmia requiring treatment
Arryhthmia | Postoperative sixth week
  Number of participants with new onset arryhthmia requiring treatment
Death | Postoperative first day
  Number of participants with mortality
Death | Postoperative sixth week
  Number of participants with mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University Dr. Rıdvan Ege Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memtsoudis SG, Sun X, Chiu YL, Stundner O, Liu SS, Banerjee S, Mazumdar M, Sharrock NE. Perioperative comparative effectiveness of anesthetic technique in orthopedic patients. Anesthesiology. 2013 May;118(5):1046-58. doi: 10.1097/ALN.0b013e318286061d. PMID 23612126
- [Background] Stundner O, Chiu YL, Sun X, Mazumdar M, Fleischut P, Poultsides L, Gerner P, Fritsch G, Memtsoudis SG. Comparative perioperative outcomes associated with neuraxial versus general anesthesia for simultaneous bilateral total knee arthroplasty. Reg Anesth Pain Med. 2012 Nov-Dec;37(6):638-44. doi: 10.1097/AAP.0b013e31826e1494. PMID 23080348